CLINICAL TRIAL: NCT04077034
Title: A Randomized, Parallel, Double Blind, Placebo Controlled Clinical Study Evaluating the Effect of Probiotic Formula on Immune System in Preschool Children
Brief Title: Effect of Probiotic Formula DE111® on Immune System in Preschool Children
Acronym: IMMUNOFORM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Deerland Enzymes (Industry)
Collaborators: Vizera d.o.o. (Industry); University of Ljubljana (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: IMMUNO-01
Record Dates: First submitted 2019-08-26; First posted 2019-09-04 (Actual); Last update posted 2019-09-04 (Actual); Status verified 2019-08

CONDITIONS: Immune System Support

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group (Experimental): Probiotic DE111®
  Interventions: Dietary Supplement: Probiotic Formula Bacillus subtilis DE111®
- Control group (Placebo Comparator): Placebo
  Interventions: Dietary Supplement: Placebo comparator

INTERVENTIONS:
Dietary Supplement: Probiotic Formula Bacillus subtilis DE111® — Probiotic Formula Bacillus subtilis DE111®, 1 billion colony forming units (CFU) per day for 8 weeks
  Arms: Experimental group
Dietary Supplement: Placebo comparator — Placebo comparator, once a day for 8 weeks
  Arms: Control group

SUMMARY:
Healthy preschool children will be recruited, gastrointestinal infection and respiratory infection symptoms will be followed during the 8-week treatment and 4-week follow-up period, to evaluate the effect of the used probiotic formula on immune system in comparison to the group using placebo.

ELIGIBILITY:
Inclusion Criteria:

* signed informed consent by at least one parent or legal guardian
* children aged 2 to 6 years
* attending or about to start attending day-care

Exclusion Criteria:

* body weight at birth <2500g
* gestational age <37 weeks
* severe chronic illness
* regular use of medication
* immunodeficiency
* parent or legal guardian not able to understand and comply with requirements of the study

Ages: 2 Years to 6 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 102 (Actual)
Dates: Start 2019-04-02 (Actual); Primary Completion 2019-08-12 (Actual); Study Completion 2019-08-12 (Actual)

PRIMARY OUTCOMES:
The incidence of gastrointestinal and/or respiratory infections for experimental group compared to control group | 12-week study period (consisting of 8-week treatment plus 4-week follow-up)
  Number of participants with at least one occurrence of gastrointestinal and/or respiratory infections during 12-week study period in the experimental group compared to control group.
The incidence of adverse events occuring in the experimental group compared to control group | 12-week study period (consisting of 8-week treatment plus 4-week follow-up)
  Number of participants with treatment related adverse events during 12-week study period for both, experimental and control group.

CONTACTS AND LOCATIONS:
Overall Officials: Lilijana Kocijancic Besednjak, MD, PhD, Principal Investigator — Health Center Nova Gorica
Locations (5):
- Slovenia (5):
  - Health center Laško, Laško
  - Pediatrija Krebs, Maribor
  - Pediatrinja d.o.o., Maribor
  - Zasebna otroska in solska ambulanta, Maribor
  - Health Center Nova Gorica, Šempeter pri Gorici

IPD SHARING:
Plan to Share IPD: No